CLINICAL TRIAL: NCT05973929
Title: Clinical and Radiological Evaluation of Movement Disorders in Multiple Sclerosis Patients.
Brief Title: Movement Disorders in Multiple Sclerosis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Hassan Meshref, Neurology physician, Al-Azhar University
Other Study IDs: Neuro-Med._0000044
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis; Movement Disorders
Keywords: Multiple sclerosis; Movement Disorders
MeSH Terms: conditions — Multiple Sclerosis; Movement Disorders | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis patients with movement disorders.: A randomized cross-sectional study will be conducted on diagnosed multiple sclerosis patients who were diagnosed according to McDonald criteria of MS 2017 (Thompson et al. 2018).
  We will study the prevalence of movement disorders in M.S patients, clinical type of movement disorder and the MRI findings. Data collected from patients admitted or following at Al-Azhar university hospitals at Al-Hussein and El-Sayed Galal hospitals. The included eligible patients should fulfil the following inclusion criteria:
  i. Full clinical history and neurological assessment. ii. Detailed multiple sclerosis history according to MS unit history sheet. iii. Detailed history of movement disorder which include clinical type of movement disorder and medication taken (or not).
  iv. MRI Brain and spine of the included patient will be photographed.
  Interventions: Other: Screen for movement disorder and correlates it with MRI findings.

INTERVENTIONS:
Other: Screen for movement disorder and correlates it with MRI findings. — * To determine the prevalence of movement disorders in MS patients.
  * To know the clinical type of movement disorders occurring with multiple sclerosis patients and the MRI finding of those patients.
  * To find the correlation between the movement disorder and the different types of MS.

SUMMARY:
The aim of this study is to determine the prevalence of movement disorders in MS patients.

Also,To know the clinical type of movement disorders occurring with multiple sclerosis patients and the MRI finding of those patients. Moreover, to find the correlation between the movement disorder and the different types of MS.

DETAILED DESCRIPTION:
A randomized cross-sectional study will be conducted on diagnosed multiple sclerosis patients who were diagnosed according to McDonald criteria of MS 2017 (Thompson et al. 2018).

The investigators will study the prevalence of movement disorders in M.S patients, clinical type of movement disorder and the MRI findings. Data collected from patients admitted or following at Al-Azhar university hospitals at Al-Hussein and El-Sayed Galal hospitals. The included eligible patients should fulfil the following inclusion criteria:

i. Full clinical history and neurological assessment. ii. Detailed multiple sclerosis history according to MS unit history sheet. iii. Detailed history of movement disorder which include clinical type of movement disorder and medication taken (or not).

iv. MRI Brain and spine of the included patient will be photographed.

Exclusion criteria:

1. Patients with multiple sclerosis mimics which can cause movement disorders e.g., systemic disease or overlap syndromes including systemic lupus, vasculitis, hepatic failure, renal failure, hyperthyroidism, electrolyte disturbances, Behcet's disease or CNS infection.
2. patients with primary movement disorders or related to other neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

- We will study the prevalence of movement disorders in M.S patients, clinical type of movement disorder and the MRI findings. Data collected from patients admitted or following at Al-Azhar university hospitals at Al-Hussein and El-Sayed Galal hospitals. The included eligible patients should fulfil the following inclusion criteria: i. Full clinical history and neurological assessment. ii. Detailed multiple sclerosis history according to MS unit history sheet. iii. Detailed history of movement disorder which include clinical type of movement disorder and medication taken (or not).

iv. MRI Brain and spine of the included patient will be photographed.

Exclusion Criteria:

- 1-Patients with multiple sclerosis mimics which can cause movement disorders e.g., systemic disease or overlap syndromes including systemic lupus, vasculitis, hepatic failure, renal failure, hyperthyroidism, electrolyte disturbances, Behcet's disease or CNS infection.

2-patients with primary movement disorders or related to other neurodegenerative diseases.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A randomized cross-sectional study will be conducted on diagnosed multiple sclerosis patients who were diagnosed according to McDonald criteria of MS 2017.
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-03-21 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence of movement disorders in MS patients. | Through study completion, an average of 1.5 year
  To know the percentage of occurance of movement disorders in MS patients.
know the clinical type of movement disorders occurring with multiple sclerosis patients and the MRI finding of those patients. | Through study completion, an average of 1.5 year
  To know the specific semiology for each movement disorder.
find the correlation between the movement disorder and the different types of MS. | Through study completion, an average of 1.5 year
  To know if there is a correlation between the movement disorder and the different types of MS.

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Mahmoud Hassan Meshref, Cairo, Select A State Or Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abboud H, Yu XX, Knusel K, Fernandez HH, Cohen JA. Movement disorders in early MS and related diseases: A prospective observational study. Neurol Clin Pract. 2019 Feb;9(1):24-31. doi: 10.1212/CPJ.0000000000000560. PMID 30859004
- [Result] Calabresi PA. Diagnosis and management of multiple sclerosis. Am Fam Physician. 2004 Nov 15;70(10):1935-44. PMID 15571060
- [Result] Cameron MH, Nilsagard Y. Balance, gait, and falls in multiple sclerosis. Handb Clin Neurol. 2018;159:237-250. doi: 10.1016/B978-0-444-63916-5.00015-X. PMID 30482317
- [Result] Dendrou CA, Fugger L, Friese MA. Immunopathology of multiple sclerosis. Nat Rev Immunol. 2015 Sep 15;15(9):545-58. doi: 10.1038/nri3871. Epub 2015 Aug 7. PMID 26250739
- [Result] Deuschl G. Movement disorders in multiple sclerosis and their treatment. Neurodegener Dis Manag. 2016 Dec;6(6s):31-35. doi: 10.2217/nmt-2016-0053. PMID 27874491
- [Result] Fragoso YD, Araujo MG, Branco NL. Kinesigenic paroxysmal hemidyskinesia as the initial presentation of multiple sclerosis. MedGenMed. 2006 Oct 4;8(4):3. PMID 17415286
- [Result] Kobelt G, Thompson A, Berg J, Gannedahl M, Eriksson J; MSCOI Study Group; European Multiple Sclerosis Platform. New insights into the burden and costs of multiple sclerosis in Europe. Mult Scler. 2017 Jul;23(8):1123-1136. doi: 10.1177/1352458517694432. Epub 2017 Feb 1. PMID 28273775
- [Result] Mehanna R, Jankovic J. Movement disorders in multiple sclerosis and other demyelinating diseases. J Neurol Sci. 2013 May 15;328(1-2):1-8. doi: 10.1016/j.jns.2013.02.007. Epub 2013 Mar 19. PMID 23522528
- [Result] Nociti V, Bentivoglio AR, Frisullo G, Fasano A, Soleti F, Iorio R, Loria G, Patanella AK, Marti A, Tartaglione T, Tonali PA, Batocchi AP. Movement disorders in multiple sclerosis: Causal or coincidental association? Mult Scler. 2008 Nov;14(9):1284-7. doi: 10.1177/1352458508094883. Epub 2008 Sep 3. PMID 18768580
- [Result] Oakes PK, Srivatsal SR, Davis MY, Samii A. Movement disorders in multiple sclerosis. Phys Med Rehabil Clin N Am. 2013 Nov;24(4):639-51. doi: 10.1016/j.pmr.2013.06.003. Epub 2013 Aug 27. PMID 24314682
- [Result] Suarez-Cedeno G, Mehanna R. Movement Disorders in Multiple Sclerosis and Other Demyelinating Diseases: A Retrospective Review From a Tertiary Academic Center. Neurologist. 2021 Sep 7;26(5):161-166. doi: 10.1097/NRL.0000000000000333. PMID 34491930
- [Result] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Result] GBD 2016 Multiple Sclerosis Collaborators. Global, regional, and national burden of multiple sclerosis 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 Mar;18(3):269-285. doi: 10.1016/S1474-4422(18)30443-5. Epub 2019 Jan 21. PMID 30679040
- [Result] Waubant E, Alize P, Tourbah A, Agid Y. Paroxysmal dystonia (tonic spasm) in multiple sclerosis. Neurology. 2001 Dec 26;57(12):2320-1. doi: 10.1212/wnl.57.12.2320. No abstract available. PMID 11756623